CLINICAL TRIAL: NCT05971394
Title: A Prospective, Multicentre, Single Arm Clinical Trial to Assess the Safety and Effectiveness of Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™) in Treating Patients With Infrapopliteal Arterial Stenosis or Occlusive Disease
Brief Title: IBS Titan™ Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotyx Medical (Shenzhen) Co., Ltd. (Industry)
Collaborators: VascuScience GmbH (Unknown); Mediolanum Cardio Research Srl (Unknown); Euroimage Research Srl (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTK-01
Record Dates: First submitted 2023-07-15; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Infrapopliteal Lesions; Critical Limb Ischemia
Keywords: BTK; below-the-knee; Infrapopliteal lesions
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBS Titan (Experimental): Subjects treated with IBS Titan™.Participants will be included in this arm.
  Interventions: Device: Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™)

INTERVENTIONS:
Device: Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™) — Subjects in this arm will be treated with Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™)

SUMMARY:
The goal of this prospective, multicentre, single arm clinical trial is to assess the safety and effectiveness of Sirolimus-eluting Iron Bioresorbable Peripheral Scaffold System (IBS Titan™) in treating patients with infrapopliteal arterial stenosis or occlusive disease. 100 participants will be implanted with IBS Titan™, and be followed up for 1-month, 6-month and 12-month after discharge.

ELIGIBILITY:
Inclusion Criteria:

• General criteria

1. Subject between 18 and 85 years old.
2. Subject who can understand the purpose of the trial, voluntarily participate in, and sign the informed consent form, and who are willing to participate until the 12 months follow-up.
3. Subject has symptomatic Critical Limb Ischemia, Rutherford category 3-5.
4. Subject requires primary treatment of de novo infrapopliteal lesions.

   • Angiographic criteria
5. Target lesion stenosis ≥ 70% or occlusion in no more than two infrapopliteal arteries.
6. The distal margin of the target lesion must be located ≥ 10 cm proximal to the proximal margin of the ankle mortise.
7. The target lesion must be located in the proximal 2/3 of native infrapopliteal vessels, length is ≤ 200mm, with vessel diameter of 2.5-4 mm.
8. Only two infrapopliteal vessels are allowed to be treated at the same time.
9. A maximum of two stents can be deployed at one target vessel.
10. There must be at least one unimpaired artery (< 30% stenosis) to the ankle.

Exclusion Criteria:

• General criteria：

1. Severe renal insufficiency, hepatic dysfunction (Cr > 2 times normal limit or renal dialysis, ALT or AST > 5 times normal limit).
2. Major amputation before index procedure or plan for major amputation.
3. Any coagulation disorder.
4. Lower extremity arteries surgery or thrombolytic therapy in the ipsilateral extremity in the past 6 weeks.
5. Stroke within 3 months, or stroke with severe hemiplegia and aphasia sequelae more than 3 months before inclusion in the study.
6. Acute myocardial infarction or acute ischemia within 30 days before inclusion in the study.
7. Thromboangiitis obliterans (Buerger's disease).
8. Any previous treatment with drug eluting balloon or drug eluting stent within 90 days before inclusion.
9. Any surgery in target vessel before index procedure.
10. Volume reduction operation in target vessel before inclusion.
11. Subject known to be allergic to aspirin, heparin, clopidogrel, Polylactic acid, iron, zinc and its degradation products, contrast agents, sirolimus, etc., and those who cannot tolerate postoperative dual anti-platelet therapy.
12. Subject with a history of iron overload or iron disorders related diseases, such as hereditary hemochromatosis, etc.
13. Subject is currently participating in another clinical trial that has not yet completed its primary endpoint.
14. Women of child-bearing potential not using an effective contraception; pregnant or lactating women.
15. Subject is not suitable to participate in the trial as per investigators discretion.
16. Life expectancy ≤ 12 months as per investigators judgement.

    • Angiographic criteria
17. The inflow tract (including ipsilateral iliac artery, femoral artery, popliteal artery) has lumen stenosis >30% with or without intervention.
18. The inflow tract (including ipsilateral iliac artery, femoral artery, popliteal artery) has > 150 mm stenosis or occlusion before treatment.
19. Significant stenosis (≥50% stenosis) of the arterial outflow tract perfused by the target vessel.
20. In-stent restenosis in any lower extremity artery.
21. Thrombosis in target vessel, or acute thrombosis requiring thrombolysis and thrombectomy.
22. Guide wire cannot pass target lesion.
23. Angiography suggests intraoperative thromboendarterectomy, percutaneous transluminal rotational atherectomy or laser therapy are needed.
24. Aneurysm of lower extremity artery in the ipsilateral leg.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from Primary Efficacy Failure | 6 months
  Defined as freedom from the composite of total occlusion of target lesion and clinically driven target lesion revascularization (CD-TLR), and freedom from major amputation.

SECONDARY OUTCOMES:
Major adverse event (MAE) | 1 month, 6 months, 12 months
  Defined as a composite of all-cause mortality, CD-TLR and major amputation of target limb.
Rate of Device success | Immediately post-procedure
  Stent level analysis, based on single stent. Defined as the achievement of successful delivery, deployment of stent at the intended infrapopliteal target site(s) and successful withdrawal of the delivery catheter.
Rate of Technical success | Immediately post-procedure
  Defined as the restoration of blood flow in the target vessel and angiogram indicates the residual stenosis <30%.
Rate of Procedural success | Immediately post-procedure
  Defined as the combination of technical success, device success, and absence of procedural complications.
Incidence of Target lesion restenosis | 1 month, 6 months, 12 months
  Defined as peak systolic velocity ratio (PSVR) >2.4 by DUS.
Change in ankle-brachial index (ABI) compared to baseline (before treatment) | 1 month, 6 months, 12 months
  Change in Ankle Brachial Index (ABI) from pre-procedure. Larger values mean a better outcome. The ABI is the systolic pressure at the ankle, divided by the systolic pressure at the arm.
Change in Rutherford Category compared to baseline (before treatment) | 1 month, 6 months, 12 months
  Categories and Clinical Description (higher scores mean a worse outcome):
  Category 0 = Asymptomatic, no hemodynamically significant occlusive disease, Category 1 = Mild claudication, Category 2 = Moderate claudication, Category 3 = Severe claudication, Category 4 = Ischemic rest pain, Category 5 = Minor tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, Category 6 = Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided